CLINICAL TRIAL: NCT02424240
Title: The Emerging Role of Serum IGF-I/IGFBP-3 Ratio in the Diagnosis of Children With Growth Hormone Deficiency
Brief Title: Growth Hormone (GH) Deficiency & Insulin Like Growth Factor 1 (IGF-I)/ Insulin Like Growth Factor Binding Protein 3 (IGFBP-3) Ratio
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Ayman Zayed, M.D., MSc, FACE, FACP, Ayman Zayed, University of Jordan
Other Study IDs: Endo-Ayman-789
Record Dates: First submitted 2015-04-18; First posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Diagnosis of GHD With IGF-I/IGFBP-3 Ratio

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IGF-I/ IGFBP-3 ratio group
  Interventions: Other: IGF-1/IGFBP-3 ratio
- IGF-1 and IGFBP-3

INTERVENTIONS:
Other: IGF-1/IGFBP-3 ratio — IGF-1/IGFBP-3 ratio for the diagnosis of GHD Vs. IGF-1, IGFBP-3 and IGF-1 & IGFBP-3 combination
  Groups: IGF-I/ IGFBP-3 ratio group

SUMMARY:
A 35-month cross-sectional observational study was conducted at an outpatient university hospital in Amman, Jordan. We obtained a comprehensive medical and laboratory evaluation for 134 short-statured children (64 boys and 70 girls, aged 4-16 years). Complete and partial growth hormone deficincy (GHD) were defined as peak forwth hormone (GH) response of 5 and 7 ng/ml [IRMA/ DiaSorin®], respectively in both clonidine stimulation and insulin tolerance tests. Serum IGF-I, IGFBP-3 and IGF-I/IGFBP-3 ratio were determined for all participants.

ELIGIBILITY:
Inclusion Criteria:

* children presented to Jordan Univeristy Hospital (JUH) outpatient endocrinology clinic for the evaluation of short stature (SS)

Exclusion Criteria:

(i) their parents could not provide written consent for them; (ii) they were lost to follow up; (iii) they could not perform clonidine stimulation tests (CST) or insulin tolerance test (ITT) due to a medical contraindication (e.g. cardiac disorder, seizure disorder); (iv) they had received GH therapy in the past; (v) they were known to have pituitary diseases, hypothyroidism, hypogonadism or discovered to have panhypopituitarism or (vi) they have malnutrition, diabetes mellitus, liver disease, or other chronic illnesses.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 192 children presented to JUH outpatient endocrinology clinic for the evaluation of short stature (SS). The target population of our study was male and female children, aged 4-16 years, with short stature.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2011-05; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Serum IGF-1/IGFBP-3 ratio | 33 months